CLINICAL TRIAL: NCT00713154
Title: A Phase II, Double-Blind Placebo-Controlled, Parallel Group Study of the Safety and Preliminary Efficacy of MTS-01, for the Prevention of Alopecia Induced by Whole Brain Radiotherapy
Brief Title: Safety and Preliminary Efficacy Study of MTS-01 for the Prevention of Alopecia Induced by WHole Brain Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Major planned study protocol modifications
Sponsor: Mitos Pharmaceuticals (Industry)
Responsible Party: Louis Habash/ President and CEO, Mitos Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Mito 02-02
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Alopecia
Keywords: Radiotherapy; induced
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo
- 2 (Active Comparator): Control Group
  Interventions: Drug: MTS-01

INTERVENTIONS:
Drug: MTS-01 — MTS-01 7% gel in 100 ml tubes, two 100 ml tubes prior to each radiation treatment
  Arms: 2
Drug: Placebo — Placebo gel in 100 ml tube, two 100 ml tubes prior to each radiation treatment
  Arms: 1

SUMMARY:
The purpose of this study is to determine if MTS-01 is effective in preventing radiotherapy-induced hair loss in patients receiving whole brain radiotherapy

DETAILED DESCRIPTION:
Hair loss (alopecia) occurs commonly as a result of external beam radiotherapy to the brain, and contributes to the social isolation and distress of patients with cancer. MTS-01 is a topical gel formulation that can be applied to the scalp during delivery of radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* is >/= 18 years of age
* Has metastatic cancer to the brain for which palliative or prophylactic whole brain radiotherapy is recommended. A histological diagnosis of cancer will be required, however, a biopsy of the brain metastases will not be required
* Can understand and sign the IRB/IEC approved informed consent, can communicate with the Investigator, and can understand with the requirements of the protocol
* has signed the HIPAA authorization

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Investigator assessment of hair loss using a 10 point scale | up to 12 weeks

SECONDARY OUTCOMES:
A time to event analysis of the hair loss | up to 12 weeks